CLINICAL TRIAL: NCT05519215
Title: A Multi-Center Evaluation of the ECHELON™ 3000 (Next Generation Powered Stapler) in General Abdominal and Thoracic Lung Resection Procedures
Brief Title: A Study of ECHELON 3000 (Next Generation Powered Stapler) in General Abdominal and Thoracic Lung Resection Procedures
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC202103; ESC202103 (Other: Ethicon, Inc.)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Sleeve Gastrectomy (LSG); Thoracic Lung Resection Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ECHELON 3000 Stapler: This prospective study will include the participants who plan to have a laparoscopic sleeve gastrectomy (LSG) or lung resection surgical procedure and collect clinical data in a post-market setting. Investigators will perform each procedure using the device in compliance with their standard surgical approach and the ECHELON 3000 Stapler and reloads instructions for use (IFU).
  Interventions: Device: ECHELON 3000 Stapler

INTERVENTIONS:
Device: ECHELON 3000 Stapler — There is no intervention, beyond necessary clinical care, in this study. Echelon 3000 Stapler is used for transection and resection in LSG or lung surgical procedure per its IFU.

SUMMARY:
The purpose of this study is to assess the safety and performance of the ECHELON 3000 Stapler (next generation powered stapler) and reload system in participants undergoing laparoscopic sleeve gastrectomy or lung resection procedures (Video-Assisted Thoracoscopic [ATS] or open approach).

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric participants satisfying the following criteria will be considered eligible for enrollment in this study (procedures may be performed with or without a robot): Primary procedure where the ECHELON 3000 Stapler and reload system is planned to be used for tissue transection per the instructions for use (IFU) in either of the following, a) Laparoscopic Sleeve Gastrectomy; b) Lung resection procedures (VATS or open)
* Adult participants- Willingness to give consent and comply with all study-related evaluations and visit schedule
* Pediatric participants- The participant's parent/legal guardian must be willing to give permission for the participant to participate in the study and provide documented informed consent for the participants. In addition, assent must be obtained from pediatric participant who possess the intellectual and emotional ability to comprehend the concepts involved in the study. If the pediatric participant is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the study), the parent/legal guardian's documented informed consent for the participant will be acceptable for the participant to be included in the study

Exclusion Criteria:

* Physical or psychological condition which would impair study participation
* Procedure is a revision/reoperation for the same indication or same anatomical location
* A procedure where surgical stapling is contraindicated
* Concurrent treatment with medications that the investigator deems could have influence on wound healing
* Enrollment in a concurrent interventional clinical study that could impact the study endpoints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who plan to have a laparoscopic sleeve gastrectomy (LSG) or lung resection surgical procedure will be included.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Select Device-related Serious Adverse Events (SAEs) | 30 days post procedure
  An adverse event (AE) is defined as any untoward medical occurrence, regardless of its relationship to study device or study procedure. An untoward medical occurrence includes any new, undesirable medical experience or worsening of pre-existing condition, which occurs throughout the duration of the clinical study. SAE is defined as an AE that results in any of the following: death; a life-threatening illness or injury; a permanent impairment of a body structure or body function; hospitalization or prolongation of existing hospitalization; medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or body function; chronic disease; fetal distress, fetal death, or a congenital physical or mental impairment or birth defect. The device-related SAEs that will be captured are infection or symptoms of infection, bleeding, gastric leak (laparoscopic sleeve gastrectomy [LSG] only), and postoperative air leak (lung resection only).

SECONDARY OUTCOMES:
Number of Participants with All Device-related, Procedure-related Adverse Events (AEs) | 30 days post-procedure
  An AE is defined as any untoward medical occurrence, regardless of its relationship to the study device or the study procedure. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition, which occurs throughout the duration of the clinical study.
Number of Participants with All Device-related, Procedure-related SAEs | 30 days post-procedure
  An AE is defined as any untoward medical occurrence, regardless of its relationship to the study device or the study procedure. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition, which occurs throughout the duration of the clinical study. A SAE is defined as an AE that results in any of the following: death; a life-threatening illness or injury; a permanent impairment of a body structure or a body function; hospitalization or prolongation of existing hospitalization; medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function; chronic disease; fetal distress, fetal death, or a congenital physical or mental impairment or birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Endo-Surgery Clinical Trial, Study Director — Ethicon Endo-Surgery
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Emory Cardiothoracic Surgery, Atlanta, Georgia
  - Henry Ford Health Center, Detroit, Michigan
  - Ascension Providence Hospital, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Bariatric Medical Institute of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Background] Qiu B, Yan W, Chen K, Fu X, Hu J, Gao S, Knippenberg S, Schwiers M, Kassis E, Yang T. A multi-center evaluation of a powered surgical stapler in video-assisted thoracoscopic lung resection procedures in China. J Thorac Dis. 2016 May;8(5):1007-13. doi: 10.21037/jtd.2016.03.88. PMID 27162678
- [Background] Fegelman E, Knippenberg S, Schwiers M, Stefanidis D, Gersin KS, Scott JD, Fernandez AZ. Evaluation of a Powered Stapler System with Gripping Surface Technology on Surgical Interventions Required During Laparoscopic Sleeve Gastrectomy. J Laparoendosc Adv Surg Tech A. 2017 May;27(5):489-494. doi: 10.1089/lap.2016.0513. Epub 2016 Dec 19. PMID 27991838